CLINICAL TRIAL: NCT05895539
Title: The Design, Implementation, and Impact of Automated Patient-reported Outcome Data Collection and Adverse Event Surveillance Tool on Treatment Continuation: an Iterative Plan-Do-Study-Act (PDSA) Approach
Brief Title: Evaluating Treatment Continuation in Telehealth Patients Receiving an Automated Patient-Reported Outcome Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-12-196-599
Record Dates: First submitted 2023-05-08; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Internet-based Intervention; Web-based Intervention; Online Intervention; Erectile Dysfunction; Telemedicine
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Did not receive the tool
- Intervention (Experimental): Did receive the tool
  Interventions: Other: An automated patient-reported outcome data collection and adverse event surveillance tool

INTERVENTIONS:
Other: An automated patient-reported outcome data collection and adverse event surveillance tool — Patients received a short prompt to provide information on treatment satisfaction and side effects
  Arms: Intervention

SUMMARY:
Engaging patients through integration of patient-reported outcome measures in routine clinical care can improve the patient experience and provide a systematic way to collect adverse event (AE) data. Collecting these data on a large scale can inform new solutions to longstanding barriers to successful treatment such as medication non-adherence.

This study evaluated whether implementing a patient-reported outcome data collection and AE surveillance tool would result in greater treatment continuation for patients receiving care on a telehealth platform. We evaluated how this data collection and surveillance tool - a short prompt for patients to provide information on treatment satisfaction and side effects - impacted the outcome of interest, treatment continuation. We tested two cycles in n=2,000 patients receiving care for erectile dysfunction on a telehealth platform using a randomized control experimental design and accounted for incidents where true randomization was not possible during implementation. The first cycle tested the tool alone, while the second cycle tested the tool in conjunction with a messaging template system that provided standardized side effect counseling.

ELIGIBILITY:
Inclusion Criteria:

* Male patients living in the US, who were diagnosed with erectile dysfunction by a telehealth provider, and who were prescribed phosphodiesterase-5 (PDE-5) inhibitors as treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Odds of refilling prescription and percent of patients who refilled prescription for patients with an initial auto-refill plan of 1 month | 91 days
  Odds of refilling prescription (logistic regression); percent of patients who refilled prescription (log rank test from Kaplan Meier curve)
Odds of refilling prescription and percent of patients who refilled prescription for patients with an initial auto-refill plan of 3 months | 123 days
  Odds of refilling prescription (logistic regression); percent of patients who refilled prescription (log rank test from Kaplan Meier curve)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Broffman, PhD, Study Director — Ro
Locations (1):
- Ro HQ, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning to share IPD at this time, due to concerns around patient privacy.

REFERENCES:
- [Derived] Zhou MS, Jain T, Hardy N, Perez-Segura A, Hickman J, Leopold L, Qualliotine K, Yedidi RS, Whetsell M, Broffman L. The design, implementation, and impact of an automated patient-reported outcome data collection and adverse event surveillance tool: a randomized trial. BMC Health Serv Res. 2023 Nov 20;23(1):1277. doi: 10.1186/s12913-023-10231-1. PMID 37986191